CLINICAL TRIAL: NCT06199063
Title: Comparison of Muscle Energy Techniques and Self-Stretching in Individuals With Nonspecific Neck Pain
Brief Title: Muscle Energy Techniques and Self-Stretching in Nonspecific Neck Pain
Acronym: METSS-NP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Ferruh Taşpınar, Study Director, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NeckPain-METSS-35
Record Dates: First submitted 2023-11-30; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Nonspecific Neck Pain; Exercise
Keywords: Neck Pain; Muscle Stretching Exercise; Electromyography; Range of Motion; Pain Threshold
MeSH Terms: conditions — Motor Activity; Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Stretching Exercises Group (SSEG) (Experimental): Self-stretching (SS) is defined as stretching applied by the individual to himself/herself. For this application, firstly the painful area was determined, and stretching was applied to the muscle with pain. Firstly, the participant stood with his/her arm free on the side to be stretched and lateral flexed his/her head. With his/her other hand, he/she applied 10 seconds of stretching in the direction of lateral flexion, a 10-second rest period was given between each stretching, and this method was performed with a total of 10 repetitions.
  Interventions: Other: Self-Streching Exercises
- Post-Isometric Relaxation Exercises Group (PIREG) (Experimental): Post-isometric relaxation (PIR) was performed by a physiotherapist in a supine position. The physiotherapist sat on the head side of the patient. The painful side was determined, and the physiotherapist fixed the head with his/her hand and performed 50% voluntary isometric contraction of the painful muscle for 10 seconds. Then, the physiotherapist asked the patient to relax and stretch for 10 seconds to lateral flexion. This method was 10 repetitions with 10 seconds of rest between each repetition.
  Interventions: Other: Post-Isometric Relaxation Exercises
- Reciprocal-Inhibition Exercises Group (RIEG) (Experimental): Reciprocal inhibition (RI) was applied by a physiotherapist in a supine position. The physiotherapist sat on the head side of the patient. The painful side was determined, and the physiotherapist fixed the head with his/her hand and performed 50% voluntary isometric contraction of the antagonist of the painful muscle for 10 seconds. Then physiotherapist asked the patient to relax and stretch for 10 seconds in the lateral flexion direction. This method was 10 repetitions and there were 10 seconds of rest between each repetition.
  Interventions: Other: Reciprocal-Inhibiton Exercises

INTERVENTIONS:
Other: Self-Streching Exercises — The participants in the SSE group; received 1 session SSE with 10 repetitions, about 30 min. The assessments were applied before and after the session.
  Other Names: SSE
  Arms: Self-Stretching Exercises Group (SSEG)
Other: Post-Isometric Relaxation Exercises — The participants in the PIRE group; received 1 session PIRE with 10 repetitions, about 30 min. The assessments were applied before and after the session.
  Other Names: PIRE
  Arms: Post-Isometric Relaxation Exercises Group (PIREG)
Other: Reciprocal-Inhibiton Exercises — The participants in the RIE group; received 1 session RIE with 10 repetitions, about 30 min. The assessments were applied before and after the session.
  Other Names: RIE
  Arms: Reciprocal-Inhibition Exercises Group (RIEG)

SUMMARY:
Non-specific neck pain (NSNP) is defined as pain not associated with neurological and specific pathologies in the posterior and lateral part of the neck between the superior nuchal line and the first thoracic vertebra. Many conservative treatment modalities including different exercise techniques are used in the treatment of NSNP. Therefore, the aim of our study was to investigate the effect of these techniques.

DETAILED DESCRIPTION:
Non-specific neck pain (NSNP) is defined as pain not associated with neurological and specific pathologies (infection, fracture, inflammation, etc.) in the posterior and lateral part of the neck between the superior nuchal line and the first thoracic vertebra. Neglecting this pain can lead to muscle spasms, stiffness, and many other serious complications. Most neck pain is caused by trigger points in the cervicothoracic muscles. Trigger points cause the muscles to weaken, and neck pain with weak cervical muscles has a negative impact on a person's quality of life.

The estimated incidence of neck pain ranges from 10.4% to 21.3% each year and is affecting an increasing number of computer and office workers. Pain intensity is low in most new cases, but disabling neck pain develops in 0.6% of the population. Therefore, it is important to investigate which treatment modality is more effective in reducing neck pain and its symptoms. Some recent studies report evidence in favor of a particular type of exercise, while others report that there is no superior type or dose of exercise.

Neck pain recurs and develops within one to five years in 20% of patients and the rate of complete recovery in these cases is very low. Neck pain is the most frequently investigated musculoskeletal problem after low back pain. It is defined as non-specific neck pain due to multifactorial etiology. Many conservative treatment modalities are used in the treatment of NSNP. These include clinical exercises, medical treatments, neural therapy, manual therapy methods, massage, acupuncture, and various physical therapy modalities. Muscle energy techniques (MET) are manual therapy methods that involve soft tissue manipulation using precise and controlled, patient-initiated, isometric, and/or isotonic contractions to improve musculoskeletal function and reduce pain. MET can be used to mobilize a joint with a limited range of motion, lengthen a spastic or shortened muscle, reduce local edema, and strengthen a physiologically weak muscle or muscle group.

Post-isometric relaxation (PIR) is defined as a reduction in the tone of the agonist muscle after an isometric contraction. This technique aims to reduce muscle tension by regulating muscle function and is used to mobilize the restricted joint, reduce edema, and lengthen and strengthen muscles in both subacute and chronic conditions. Studies have also used PIR for neck pain.

The muscle spindle is one of the sensory receptors in skeletal muscle. Its function is to provide proprioceptive information to the cerebral cortex. As the muscle lengthens, the muscle spindle is activated, and a reflex contraction of the agonist muscle and relaxation of the antagonist muscle occurs. This process is known as reciprocal inhibition (RI). Studies using the RI technique in people with neck pain were found. However, no studies were found in people with non-specific neck pain.

Stretching is a general term describing a therapeutic maneuver used to increase the extensibility of soft tissues. Self-stretching (SS) is the self-application of this technique. Studies comparing the effects of MET with different treatment modalities in people with non-specific neck pain were identified in the literature. These trials found similar effects and varying degrees of superiority in reducing pain intensity and increasing range of motion (ROM). In the literature, studies have compared stretching with MET in people with neck pain or compared MET with different treatment methods and examined their effects on variables such as pain and ROM. However, no study was found that compared different METs and self-training in individuals with NSNP and investigated the immediate effect of EMG. Therefore, the aim of our study was to investigate the effect of these techniques. It was thought that the information obtained as a result of the study would guide the creation and development of rehabilitation programs.

The hypotheses of the study are as follows:

Hypothesis 1: The PIR technique applied to individuals with NSNP has a positive effect on pain intensity, pressure pain threshold, range of motion, and muscle activation.

Hypothesis 2: The RI technique applied to individuals with NSNP has a positive effect on pain intensity, pressure pain threshold, range of motion, and muscle activation.

Hypothesis 3: SS technique applied to individuals with NSNP has a positive effect on pain intensity, pressure pain threshold, range of motion, and muscle activation.

Hypothesis 4: Muscle energy techniques applied to individuals with NSNP have more positive effects on pain intensity, pressure pain threshold, range of motion and muscle activation than SS technique.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Being a volunteer to participate into the study
* Not having diagnosed orthopedic and neurological problems
* Having Neck pain for at least four months

Exclusion Criteria:

* Having diagnosed with active infectious pathology
* Having cervical spine fracture/previous cervical or thoracic surgery
* Having a history of severe trauma to the cervical spine
* Having a history of malignant tumors
* Having diagnosed with structural deformity
* Being used of a medical orthopaedic prosthesis
* Having a pacemaker
* Having diagnosed with disc prolapse

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-02-04 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain Severity | Before and up to 4 weeks
  Pain severity was assessed using the Visual Analogue Scale (VAS). The VAS is a subjective pain scale in which the intensity of pain is rated 0-10 cm on a horizontal line. "0" refers to "no pain, while "10" refers to worst pain.
Assessment of Pressure Pain Threshold | Before and up to 4 weeks
  The Wagner digital algometer (Wagner Instruments) was used to measure the pressure pain threshold (PPT). Trigger points in the upper trapezius and cervical paravertebral muscles were palpated and the most painful trigger points were marked as four separate points on the right and left. The algometer was placed perpendicular to the trigger points and the pressure was increased until the first moment when the patient felt pain and the probe was withdrawn with the expression "I felt it/OK". At this point, the PPT value in Newton read from the algometer was recorded in three repetitions.
Assessment of Range of Motion | Before and up to 4 weeks
  The subjects' neck ROMs were recorded in degrees by measuring the degrees of flexion, extension, lateral flexion and rotation three times with a manual goniometer while sitting upright in a chair.
Assessment of Muscle Activation | Before and up to 4 weeks
  Muscle activation was assessed with a MegaWin WBA eight-channel EMG device. Superficial EMG electrodes were placed on the upper trapezius and sternocleidomastoid muscles, right and left. A total of 4 outputs were used, 2 muscles on each side. Myoelectric signals were obtained, and muscular contraction and inhibition were assessed. Additionally, the "IC/MVIC" percentage was calculated to determine the workload on the muscle during the activity.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Taspinar, Prof. Dr., Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No